CLINICAL TRIAL: NCT02248012
Title: Everolimus and Temozolomide as 1-line Treatment in Advanced Gastroenteropancreatic Neuroendocrine Carcinoma (G3) With a Ki67 of 20-55%
Brief Title: Everolimus and Temozolomide in Advanced Gastroenteropancreatic Neuroendocrine Carcinoma (G3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Skane University Hospital (Other); Copenhagen University Hospital, Denmark (Other); Rigshospitalet, Denmark (Other); Uppsala University Hospital (Other); Aarhus University Hospital (Other); Sahlgrenska University Hospital (Other); Ullevaal University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-002524-16
Record Dates: First submitted 2014-07-24; First posted 2014-09-25 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Neuroendocrine Carcinoma
Keywords: Gastroenteropancreatic; Neuroendocrine carcinoma; Chemotherapy
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Everolimus; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus/temozolomide (Experimental): Everolimus 10 mg daily, temozolomide 150 mg/m2 for 7 days every 2 weeks.
  Interventions: Drug: Everolimus , temozolomide

INTERVENTIONS:
Drug: Everolimus , temozolomide

SUMMARY:
To study the efficacy of everolimus combined with temozolomide as first-line treatment in advanced gastroenteropancreatic neuroendocrine carcinoma with a Ki67 of 20-55%, measured as disease control rate (non-progressive disease) at 6 months.

DETAILED DESCRIPTION:
Guidelines for treating advanced gastroenteropancreatic neuroendocrine carcinomas (GEP-NECs) advocate the use of combination chemotherapy with a platinum-based chemotherapy combined with etoposide. No other regimen has consistently shown a benefit over this combination. NECs do not respond to treatments usually applied in other neuroendocrine tumours such as somatostatin analogues and interferon. In contrast to metastatic neuroendocrine tumours with a low Ki67, debulking surgery and surgery for liver metastasis is generally not recommended. Cisplatin /carboplatin and etoposide is established as standard treatment of advanced disease based on two small retrospective studies showing a response rate between 41- 67% and median survival of 15-19 months. In the current trial we propose an alternative treatment for a subgroup of patients with GEP-NEC based on new data, with the intention to improve response rates and clinical benefit rate without increasing toxicity

ELIGIBILITY:
Inclusion criteria

Histologically proven neuroendocrine carcinoma with a Ki67 of 20-55%.Primary gastroenteropancreatic tumor or cancer of unknown primary where metastases are mainly abdominalMeasurable disease according to RECIST by CT/MR

General conditions:

* >18 years;
* WHO/ECOG performance status 0-1.
* Adequate haematological, renal and hepatic functions:
* Written informed consent prior to inclusion

Prior therapy:

* No prior chemotherapy treatment for advanced disease.
* Adjuvant chemotherapy must have ended > 6 months before inclusion.

Prior or current history:

* No curatively resectable disease;
* No other serious illness or medical conditions (including: unstable angina, myocardial infarction within 6 months, unstable diabetes, immune suppression )

Concomitant treatments :

* No concomitant (or within 4 weeks before inclusion) administration of any other experimental drug;
* No other concurrent anti-cancer therapy.

Other :

* Not pregnant or breast feeding. Fertile patients must use adequate contraceptives and fertile females must have a negative pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Disease control rate | 6 months

SECONDARY OUTCOMES:
Number of patients with adverse events | During treatment + 30 days
  Especially number of patients with grade 3-4 toxicity.

OTHER OUTCOMES:
Time (months) from start of study treatment to death (survival) | Average 14 months
  Patients alive at 18 months after last patient entered into the study will be censored.

CONTACTS AND LOCATIONS:
Overall Officials: Halfdan Sorbye, MD, Principal Investigator — Haukeland Univ Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Background] Sorbye H, Strosberg J, Baudin E, Klimstra DS, Yao JC. Gastroenteropancreatic high-grade neuroendocrine carcinoma. Cancer. 2014 Sep 15;120(18):2814-23. doi: 10.1002/cncr.28721. Epub 2014 Apr 25. PMID 24771552